CLINICAL TRIAL: NCT02188576
Title: The Efficacy and Population Pharmacokinetics/ Pharmacogenomics of a Reduced Dose of Tranexamic Acid for Craniosynostosis Surgery
Brief Title: The Efficacy and Population Pharmacokinetics of Tranexamic Acid for Craniosynostosis Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Susan Goobie, Senior Assistant in Perioperative Anesthesia, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P00008434
Record Dates: First submitted 2014-07-10; First posted 2014-07-11 (Estimated); Results first posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Craniosynostosis
Keywords: Craniofacial Surgery; tranexamic acid; Antifibrinolytic
MeSH Terms: conditions — Craniosynostoses | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- high dose TXA (Experimental): High dose TXA is the intervention.
  A higher dose of tranexamic acid will be given to this arm as follows:
  50 mg/kg loading dose and 5 mg/kg/h infusion
  Interventions: Drug: high dose TXA
- Low Dose TXA (Experimental): Low dose TXA is the intervention.
  A lower dose of TXa will be given as follows:
  10 mg/kg loading dose and 5 mg/kg/h infusion
  Interventions: Drug: Low dose TXA

INTERVENTIONS:
Drug: high dose TXA
  Other Names: Tranexamic acid, Cyclokapron; Craniofacial surgery
  Arms: high dose TXA
Drug: Low dose TXA
  Other Names: Tranexamic Acid, cyclokapron,; Craniofacial surgery
  Arms: Low Dose TXA

SUMMARY:
This research study is being performed to evaluate two different doses of Tranexamic acid (TXA) in children who have craniosynostosis and have been referred to Boston Children's Hospital for corrective surgery. This surgery is associated with significant blood loss and frequently requires the transfusion of blood. TXA is a medication that reduces the amount of bleeding during surgery by improving clotting of the blood at the surgical site. TXA is an FDA-approved drug that is routinely used in infants and children undergoing major surgery including heart surgery, craniofacial surgery and scoliosis surgery. It has been shown to decrease both the amount of bleeding and the amount of blood transfusion needed. We would like to compare the different doses of TXA to see if a lower dose has the same effect on blood loss as a higher dose. We are also interested to learn why TXA seems to work better in some patients than in others. In order to study the effect of this drug we would like to give this drug to your child and measure the blood loss and the volume of blood given to your child during his/her surgery.

The research is being done at two sites; Boston Children's Hospital and Gaslini Children's Hospital in Genoa, Italy. The main study doctor from Boston Children's Hospital is Dr. Susan Goobie. The Department of Anesthesiology at Boston Children's Hospital is sponsoring this study.

We are planning to study a total of 68 infants and children from age 3 months to 6 years old scheduled for open craniosynostosis surgery at Boston Children's Hospital or Gaslini Children's Hospital.

DETAILED DESCRIPTION:
Introduction: Over 90% of open craniosynostosis surgical procedures are associated with a transfusion of blood or blood products. Goobie et. al. recently showed that tranexamic acid in a dose of 50 mg/kg/15min and 5 mg/kg/h significantly reduced blood loss and transfusion requirements as well as the overall exposure of children to donor PRBC by two thirds. However, using a moderately high dosing regimen, TXA plasma concentrations were shown to far exceed the accepted therapeutic level (by over 10 fold). No side effects of TXA were found in this study but a recent study suggests that currently recommended high to moderate TXA dosing regimens are potentially associated with neurological complications in children. Goobie et. al. developed a population pharmacokinetic model of TXA and simulated a dose response curve for this population. From this model and simulation, it appears that reducing the loading dose to 10 mg/kg/15 min followed by a 5 mg/kg/h infusion is adequate to maintain plasma concentrations above the accepted therapeutic level of 20ug/mL.

It is important to test and validate this reduced dosage scheme in a multicenter study. The hypothesis is that this reduced dosage scheme (10 mg/kg loading dose and 5 ug/kg/h) is as effective as the higher dosage scheme (50 mg/kg loading dose and 5 mg/kg/h) in decreasing blood loss and transfusion requirements in children undergoing open craniosynostosis surgery. Thus the PK/PD profile of TXA in craniosynostosis patients will be determined with genomics explored as a cause of interpatient variability in the response to tranexamic acid.

Experimental Design: With IRB approval and informed consent 68 pediatric patients aged 3 m to 6 years coming for open craniofacial surgery will be randomized in a prospective double blind fashion to either the current standard intravenous TXA dose (50mg/kg/15min and 5 mg/kg/h) or this lower TXA dose (10 mg/kg/15min and 5 mg/kg/h) until the end of surgery. A standardized anesthetic and well defined fluid, blood and blood product management protocols will be followed with improved modifications from the previously described protocol.

Data Analysis Plan: A preliminary power analysis indicated that a total sample size of 56 children (28 in randomized each group) would provide 80% statistical power to test whether the difference in average blood loss is equivalent to within 25% (ie 15 cc/kg) assuming a standard deviation of 30% ie +/- 22 ml/kg (moderate effect size = 0.68) . We plan to randomize 68 patients; 34 per group to ensure that we meet our sample size requirements while accounting for a potential 20% patient drop out.

Specific Aims:

1. Determine the efficacy of TXA (PD) in infants and children undergoing open craniofacial surgery with this lower dosage scheme.
2. Determine the population pharmacokinetics (PK) of TXA in infants and children undergoing open craniofacial surgery with this dosage scheme.
3. Determine the influence of genetics on response to TXA.
4. Attempt to better define efficacy of TXA in a direct manner using a novel and innovative approach by obtaining pre and post biological markers of fibrinolysis (as bleeding and blood loss are difficult to measure accurately and are an indirect measure of TXA efficacy of inhibition of fibrinolysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients (age range 3 months to 6 years) undergoing craniosynostosis repair, fronto-orbital advancement surgery and cranial remodeling surgery (i.e. total cavernal remodeling surgery).

Exclusion Criteria:

* Preexisting hematological abnormality (defined as a positive history of bleeding disorder or a known diagnosis of a genetic or acquired bleeding disorder)
* Preexisting coagulation defect (defined as PT, PTT or INR >1.5 times normal or a n pre-existing genetic or acquired coagulation defect))
* Preexisting hepatic, renal, vascular, ocular and/or metabolic disorder
* History of acetylsalicylate ingestion within the last 14 days.
* History of NSAIDs ingestion with 2 days of the scheduled surgery date

Ages: 3 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2014-08; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Goobie, MD, Principal Investigator — Boston Children's Hospital; Nicola Disma, MD, Principal Investigator — Gaslini Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goobie SM, Staffa SJ, Meara JG, Proctor MR, Tumolo M, Cangemi G, Disma N. High-dose versus low-dose tranexamic acid for paediatric craniosynostosis surgery: a double-blind randomised controlled non-inferiority trial. Br J Anaesth. 2020 Sep;125(3):336-345. doi: 10.1016/j.bja.2020.05.054. Epub 2020 Jun 30. PMID 32620262

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment locations were the preoperative clinics at Boston Children's Hospital (Boston, MA) and Gaslini Children's Hospital (Genoa, Italy) from 2014 to 2017.
Groups:
- High Dose TXA: High dose TXA is the intervention.
  A higher dose of tranexamic acid will be given to this arm as follows:
  50 mg/kg loading dose and 5 mg/kg/h infusion
  high dose TXA
- Low Dose TXA: Low dose TXA is the intervention.
  A lower dose of TXa will be given as follows:
  10 mg/kg loading dose and 5 mg/kg/h infusion
  Low dose TXA
Period: Overall Study
Arm/Group | High Dose TXA | Low Dose TXA
Started | 32 | 34
Completed | 32 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose TXA | Low Dose TXA | Total
Number analyzed (Participants) | 32 | 34 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32 | 34 | 66
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Inter-Quartile Range); unit: months] | 8 [4 to 13.5] | 8.5 [5 to 16] | 8.25 [4 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 19 | 21 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 32 | 34 | 66
Region of Enrollment [Number; unit: participants]
  United States | 12 | 14 | 26
  Italy | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of TXA in Childrens Having Craniosynostosis Surgery
Description: Determine the efficacy ( as measured by blood loss and blood transfusion) of TXA in infants and children undergoing open craniofacial surgery with this lower dosage scheme.
Time Frame: perioperatively from the intraoperative period to 24 hours postoperatively
Population: To determine if a tranexamic acid dose regimen of 10 mg/kg loading dose and 5 mg/kg/h maintenance dose is as effective as a higher dose regime of 50 mg/kg loading dose and 5 mg/kg/h maintenance infusion rate in reducing blood transfusion volume in pediatric craniosynostosis reconstruction surgery.
Measure: Mean (Standard Error); unit: mL/kg
Groups:
- High Dose TXA: High dose TXA is the intervention.
  A higher dose of tranexamic acid will be given to this arm as follows:
  50 mg/kg loading dose and 5 mg/kg/h infusion
  high dose TXA
  Outcome: A tranexamic acid dose regimen of 10 mg/kg loading dose and 5 mg/kg/h maintenance dose is as effective as a higher dose regime of 50 mg/kg loading dose and 5 mg/kg/h maintenance infusion rate in reducing blood loss and transfusion requirements in pediatric craniosynostosis reconstruction surgery.
- Low Dose TXA: Low dose TXA is the intervention.
  A lower dose of TXa will be given as follows:
  10 mg/kg loading dose and 5 mg/kg/h infusion
  Low dose TXA
  Outcome: A tranexamic acid dose regimen of 10 mg/kg loading dose and 5 mg/kg/h maintenance dose is as effective as a higher dose regime of 50 mg/kg loading dose and 5 mg/kg/h maintenance infusion rate in reducing blood loss and transfusion requirements in pediatric craniosynostosis reconstruction surgery.
Arm/Group | High Dose TXA | Low Dose TXA
Number analyzed (Participants) | 32 | 34
mL/kg | 23.6 (1.5) | 21.3 (1.6)

2. Secondary Outcome: Plasma Levels of TXA in Children Having Craniosynostosis Surgery
Description: Determine the plasma levels (in micrograms/mL) of TXA in infants and children undergoing open craniofacial surgery with this dosage scheme
Time Frame: up to 24h postoperatively
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | High Dose TXA | Low Dose TXA
Number analyzed (Participants) | 32 | 34
ug/mL | 50.2 (8.0) | 29.6 (7.6)

ADVERSE EVENTS:
Time Frame: while the patient was in hospital which was up to a maximum of 15 days
Description: side effects including VTE, seizures
Arm/Group | High Dose TXA | Low Dose TXA
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/34
Other Adverse Events (participants affected / at risk) | 0/32 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/76/NCT02188576/Prot_SAP_000.pdf